CLINICAL TRIAL: NCT03468608
Title: Development and Validation of a Pediatric Procedural Sedation Satisfaction Survey
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mark Crawford, Anesthesiologist-in-Chief, The Hospital for Sick Children
Other Study IDs: 1000056420
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Satisfaction
Keywords: procedural sedation; paediatric; parental satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phase 1: Instrument Development: An initial set of questionnaire items will be created based on the questionnaires noted in the literature review as well as the semi-structured interviews conducted with parents and healthcare team members in our facility.
- Phase 2: Pre-Test Evaluation: Parents and healthcare team members will be asked to comment on the quality of the draft questionnaire created in phase 1 of this study.
- Phase 3: Pilot: Parents will be asked to complete the questionnaire developed during phase 2 of this study. Upon completing the questionnaire, parents will be asked to rate the overall face validity of the tool using a 5-point Likert scale.
  Healthcare team members will be asked to rate the content validity of each item on the questionnaire.
- Phase 4: Validation: Parents will be asked to complete the questionnaire developed during phase 3 of this study.

SUMMARY:
The quality of care associated with medical procedures, such as procedural sedation, has historically been assessed from the perspective of the healthcare professional, wherein the appropriateness of the services provided and the skill with which this care was performed were considered. However, more recently, the perspectives of consumers of healthcare services (i.e. the patients) have also been sought in the form of patient satisfaction. A review of the literature shows that patient satisfaction is routinely assessed when determining the effectiveness of sedation; however, it is less frequently assessed as the primary outcome. In child-specific, validated studies, limitations are noted with respect to being validated in a language other than English and failing to encompass a variety of procedures. As a result, these validated tools are not appropriate for use with pediatric populations undergoing procedural sedation in North America, nor are these validated tools amenable to comparison with our proposed tool.

DETAILED DESCRIPTION:
Due to the central unit procedural sedation team servicing several areas of specialty, a varied patient satisfaction tool is required to ensure all concerns pertaining to sedation in each specialty are addressed, as well as allowing consistency between specialties to be examined. Therefore, the objective is to develop and validate a procedural sedation satisfaction tool for use with a variety of specialties requiring pediatric procedural sedation.

ELIGIBILITY:
Inclusion Criteria for Parents:

* child is receiving procedural sedation within the central unit at our facility
* child is aged 0-8 years

Exclusion Criteria for Parents:

* parent self-identifies as not being able to speak or read English

Inclusion Criteria for Healthcare Team Members:

* work within the central unit providing procedural sedation at our facility

Exclusion Criteria for Healthcare Team Members:

* none

Max Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parent population will be based on those receiving services within our central unit.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Parental Satisfaction with Procedural Sedation | immediately proceeding procedural sedation experience
  determined via development/validation of a parental satisfaction tool

CONTACTS AND LOCATIONS:
Overall Officials: Mark Crawford, Principal Investigator — Anesthesiologist-in-Cheif
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada